CLINICAL TRIAL: NCT05825079
Title: A Randomized, Parallel, Two Arm, Unblinded Single-center Study of the Effects of Patient-provided Feedback on Fracture Healing and Weight-bearing Status in Orthopedic Patients Undergoing Operative Fixation or Non-operative Treatment of Isolated Tibial Plateau, Pilon, and Other Ankle Fractures
Brief Title: Does Weightbearing Crutch Technology Impact Patient Compliance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: ComeBack Mobility (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-01427
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Fracture Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-Bearing Feedback Delivered to Mobile Phone (Experimental): The weight-bearing tracking system is attached to the patient's crutch and calculates how much weight is being put on the crutch. Feedback of this data can be delivered to the patient through a mobile phone application. For Arm A of the study, feedback is delivered to the patient's paired mobile phone, providing them information on how much weight they are exerting on their crutch/injured lower extremity.
  Interventions: Behavioral: Weight-Bearing Feedback; Device: Smart Crutch Tip
- No Weight-Bearing Feedback (Active Comparator): The weight-bearing tracking system is attached to the patient's crutch and calculates how much weight is being put on the crutch. For Arm B, no feedback about weight-bearing status is delivered to the patient.
  Interventions: Device: Smart Crutch Tip

INTERVENTIONS:
Behavioral: Weight-Bearing Feedback — Feedback on how much weight patients are exerting on their crutch/injured lower extremity (measured via Smart Crutch Tip) will be delivered to their mobile phones.
  Arms: Weight-Bearing Feedback Delivered to Mobile Phone
Device: Smart Crutch Tip — The device is attached to the crutch and measures how much weight-bearing load is exerted onto its axis. The device is capable of transmitting this data into the patient and physicians' user interface.

SUMMARY:
The goal of this study is to determine if weight-bearing crutch technology that delivers active feedback to patients during their treatment will impact patient compliance with physician instructions.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate in study and complete consent
* Will undergo treatment of an isolated tibial plateau, pilon, or ankle fracture and placed in a non-weightbearing status with the use of crutches at NYU.
* Have access and use of a mobile phone (exclusively iOS and/or Android devices)

Exclusion Criteria:

* Patients with concomitant TBI
* Polytrauma patients
* Pathologic fractures
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Percent (%) Change in Average Weight On Crutch from Week 2 to Week 12 | Week 2, Week 12
  Average weight put on crutch measured using the Smart Crutch Tip.

SECONDARY OUTCOMES:
Time to Recovery | Up to Week 12
  Measured as the duration of time from treatment (operative or non-operative) to recovery.
Change in Visual Analogue Scale (VAS) - Pain Score from Baseline to Week 12 | Baseline, Week 12
  Participants rate pain using a VAS ranging from 0 (no hurt) to 10 (unbearable pain). A decrease in scores indicates pain decreased during the observational period.
Percent (%) of Participants with Injury Complications | Up to Week 12
Percent (%) of Participants who Experience Nonunion/Malunion of Lower Extremity Injury | Up to Week 12
  Nonunion/malunion assessed using radiographic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A. Egol, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Kenneth.Egol@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. equests should be directed to Kenneth.Egol@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.